CLINICAL TRIAL: NCT05634811
Title: A PHASE 3, RANDOMIZED, PLACEBO-CONTROLLED, OBSERVER-BLINDED TRIAL TO EVALUATE THE SAFETY OF A 6-VALENT OspA-BASED LYME DISEASE VACCINE (VLA15) IN HEALTHY CHILDREN 5 THROUGH 17 YEARS OF AGE
Brief Title: Safety Study of a Vaccine to Help Protect Against Lyme Disease in Healthy Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: C4601012; NCT05634811 (Registry Identifier: ClinicalTrials.gov); 2025-000441-15 (EudraCT Number)
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Lyme Disease
Keywords: Borreliosis; Borrelia burgdorferi; Spirochetes; Vector-Borne Disease; Lyme Disease Vaccine; VLA15; Outer Surface Protein A (OspA); Ticks
MeSH Terms: conditions — Lyme Disease; Borrelia Infections; Vector Borne Diseases | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VLA15 (Experimental): Participants will receive 6-valent OspA-based Lyme disease vaccine (VLA15).
  Interventions: Biological: VLA15
- Normal Saline (Placebo) (Placebo Comparator): Participants will receive 0.9% sodium chloride solution for injection
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: VLA15 — 6-valent OspA-based Lyme disease vaccine
  Other Names: PF-07307405
  Arms: VLA15
Other: Normal Saline — 0.9% sodium chloride solution for injection
  Arms: Normal Saline (Placebo)

SUMMARY:
This study is to understand if the study vaccine (called VLA15) is safe in healthy children.

We are looking for children who:

* are healthy
* are age 5 through 17
* have not been diagnosed with any form of Lyme disease in the past
* have not received any vaccines for Lyme disease in the past

Lyme disease happens most often in children of this age. The study vaccine may be used potentially to help prevent Lyme disease. The goal of this study is to get more information about the safety of the study vaccine in this age group.

Participants will be in this study for about 2 years. During that time, they will receive VLA15 or placebo (sterile saltwater solution) by a "shot" in the arm. We will compare experience of children receiving VLA15 to those receiving the placebo. Participants will not know whether they get VLA15 or placebo.

Everyone participating in this study will:

* get the shots in a clinic or in a hospital office
* receive a total of 4 shots
* receive the first 3 shots within 6 months
* receive the last shot about 1 year afterwards
* need to come to the trial site for 6 planned visits; 4 of these are vaccination visits and 2 are follow-up visits. We will contact you by phone 1 time every year during the study to monitor your experience. You may have extra visits if you experience a severe reaction after a vaccine dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants at enrollment who are determined to be eligible for inclusion in the study. Participants with preexisting chronic medical conditions determined to be stable may be included.
* Participants and/or participants' parent(s)/guardian who are willing and able to comply with all scheduled visits, study procedures and lifestyle considerations for the duration of the study.

Exclusion Criteria:

* Female participants that are pregnant, breastfeeding, or have a positive urine pregnancy test at Visit 1. Sexually active females and fertile males unwilling to use contraception as per protocol.
* Any contraindication to vaccination or vaccine components, including previous anaphylactic reaction to any vaccine or vaccine-related components.
* Any diagnosis of Lyme disease within the past 3 months.
* Any history of Lyme arthritis, carditis, neuroborreliosis, or other disseminated Lyme Disease (LD), regardless of when diagnosed.
* Known tick bite within the past 4 weeks.
* Congenital or acquired immunodeficiency or other conditions or treatments associated with immunosuppression that would inhibit the ability to mount an immune response to a vaccine.
* Other medical, psychiatric condition, active suicidal ideation/behavior or lab abnormality which increases risk of study participation or, in investigator's judgment is inappropriate for the study.
* Receipt of a previous vaccination for LD.
* Treatment for LD in the 3 months prior to study intervention administration.
* Receipt of blood/plasma products or immunoglobulins within 6 months before study intervention administration through conclusion of the study.
* Receipt of systemic corticosteroids for ≥14 days within 28 days before study intervention administration. Inhaled/nebulized, intra-articular, intrabursal, or topical corticosteroids are permitted.
* Receipt of chronic systemic treatment with other known immunosuppressant medications, or radiotherapy, within 6 months before study intervention administration.
* Current use of any prohibited concomitant medication(s) or participants unwilling/unable to use a permitted concomitant medication(s).
* Participation in other studies involving investigational drugs/vaccines/devices within 28 days prior to study entry and/or during study participation (observational studies are acceptable).
* Investigator site staff, sponsor/sponsor delegates directly involved in the conduct of the study and their family members; site staff supervised by the investigator and their family members.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3549 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
The percentage of participants reporting prompted local reactions | Within 7 days following each study intervention administration
The percentage of participants reporting prompted systemic events | Within 7 days following each study intervention administration
The percentage of participants reporting adverse events (AEs) | Through 1 month following each study intervention administration
The percentage of participants reporting newly diagnosed chronic medical conditions (NDCMCs) | Through study completion, up to 24 months
The percentage of participants reporting serious adverse events (SAEs) | Through study completion, up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (65):
- United States (65):
  - UAB Child Health Research Unit (CHRU), Birmingham, Alabama
  - University of Alabama at Birmingham - School of Medicine, Birmingham, Alabama
  - Lakeview Clinical Research, Guntersville, Alabama
  - Coast Clinical Research, LLC, Bellflower, California
  - Apex Research Group LLC, Fair Oaks, California
  - New England Research Associates, Bridgeport, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Bio-Medical Research LLC, Miami, Florida
  - GCP Research, Global Clinical professionals, St. Petersburg, Florida
  - MOORE Clinical Research, Inc. d/b/a TrueBlue Clinical Research, Tampa, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Tekton Research, LLC., Chamblee, Georgia
  - ASR, LLC, Boise, Idaho
  - Clinical Research Prime, Idaho Falls, Idaho
  - Clinical Research Prime Rexburg, Rexburg, Idaho
  - University of Chicago Medical Center, Chicago, Illinois
  - AMR Clinical, El Dorado, Kansas
  - AMR Clinical, Wichita, Kansas
  - Kentucky Pediatric/ Adult Research, Bardstown, Kentucky
  - All Children Pediatrics, Louisville, Kentucky
  - MD Medical Research, Oxon Hill, Maryland
  - White Oak Pediatrics, Silver Spring, Maryland
  - Sisu BHR, Springfield, Massachusetts
  - Michigan Center of Medical Research (MICHMER), Bingham Farms, Michigan
  - Vida Clinical Studies, LLC, Dearborn Heights, Michigan
  - Great Lakes Research Institute, Southfield, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - Velocity Clinical Research, Omaha, Omaha, Nebraska
  - Hassman Research Institute, Marlton, New Jersey
  - Rutgers University, New Brunswick, New Jersey
  - IMA Clinical Research Warren, Warren Township, New Jersey
  - Velocity Clinical Research, Binghamton, Binghamton, New York
  - Buffalo Clinical and Translational Research Center, Buffalo, New York
  - Advanced Specialty Care, Commack, New York
  - Smith Allergy and Asthma Specialists, Cortland, New York
  - Stony Brook Medicine Clinical Research Center, East Setauket, New York
  - Upstate Global Health Institute, East Syracuse, New York
  - Southampton Hospital, Hampton Bays, New York
  - Smith Allergy & Asthma Specialists, Horseheads, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - DiGiovanna Institute for Medical Education & Research, North Massapequa, New York
  - Rochester Clinical Research, LLC, Rochester, New York
  - Stony Brook University, Stony Brook, New York
  - Prime Global Research, The Bronx, New York
  - Advantage Clinical Trials, The Bronx, New York
  - Velocity Clinical Research, Vestal, Vestal, New York
  - Centricity Research Columbus Ohio Multispecialty, Columbus, Ohio
  - Allegheny Health and Wellness Pavilion, Erie, Pennsylvania
  - Central Erie Primary Care, Erie, Pennsylvania
  - Preferred Primary Care Physicians, Preferred Clinical Research (Ofc 18), Pittsburgh, Pennsylvania
  - Northeast Clinical Trials Group, Scranton, Pennsylvania
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Benchmark Research, Austin, Texas
  - Benchmark Research, Fort Worth, Texas
  - Texas Health Resources, Fort Worth, Texas
  - C & R Research Services USA, Houston, Texas
  - DM Clinical Research - Kool Kids Pediatrics, Houston, Texas
  - Research Your Health, Plano, Texas
  - Sun Research Institute, San Antonio, Texas
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Pediatric Research of Charlottesville, LLC, Charlottesville, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Frontier Clinical research, Kingwood, West Virginia
  - Preston Healthcare Services, Kingwood, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4601012